CLINICAL TRIAL: NCT02560818
Title: Transcriptomes Breast, Ovarian and Leukocyte Hereditary Genes Predisposing to Breast and / or Ovarian Cancer
Acronym: CASOHAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Francois Baclesse (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CASOHAR
Record Dates: First submitted 2015-09-24; First posted 2015-09-25 (Estimated); Last update posted 2020-11-09 (Actual); Status verified 2020-11

CONDITIONS: Breast Cancer; Transcriptomes; Molecular Diagnostic; Ovarian Cancer
Keywords: splice profiles of messenger RNA
MeSH Terms: conditions — Breast Neoplasms; Ovarian Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control population : Healthy Volunteers (Active Comparator): 20 Healthy Volunteers will be recruited:
  * 10 women to recover breast tissue (from surgical waste) : populations A and C
  * 10 women to recover ovarian tissue (from surgical waste) : population B
  Interventions: Other: collection of a blood sample and breast and ovarian tissue
- Patients (Experimental): blood samples of 50 patients will be used (use of blood collection in study EXSAL N°ID-RCB 2009-A00833-54)
  Interventions: Other: use of a previous blood collection for patients

INTERVENTIONS:
Other: collection of a blood sample and breast and ovarian tissue — a blood sample and a breast and ovarian tissue sample will be collected in healthy women during their surgery (breast or ovarian surgery according to selection group :A, B or C)
  Arms: Control population : Healthy Volunteers
Other: use of a previous blood collection for patients
  Arms: Patients

SUMMARY:
This is a case-control study of molecular diagnostics.

This study requires two steps:

* The first part of the study will be conducted on a population of 20 women without breast cancer and, or ovarian family (Healthy Volunteers controls)
* The second part of the study will be conducted on a population of 50 patients predisposed to familial breast and, or ovarian cancer compared to 20 controls .

For analysis of leucocytes of the patients, a blood sample collected in a prior study (EXSAL study, ID-RCB 2009-A00833-54) will be used.

DETAILED DESCRIPTION:
This study requires two steps:

- The first part of the study will be conducted on a population of 20 women free of breast cancer and, or ovarian Family (healthy volunteers controls) and without a known family history of breast and or ovarian cancer.

Mapping the level of blood (leukocytes) and the breast tissue will be drawn for the same individual on the physiological profiles splicing of the messenger RNA of genes involved in this predisposition, targeted by high-throughput sequencing of RNA (RNASeq).

A direct comparison of RNA splicing patterns between blood and breast tissue from the same witness will detect any differences between these two tissues.

-The second part of the study will be conducted on a population of 50 patients predisposed to familial breast and, or ovarian cancer compared to 20 controls with no known family history of breast and, or ovarian cancer.

Analysis of the results will highlight potential splicing abnormalities.

ELIGIBILITY:
For Healthy Volunteers

Inclusion Criteria:

For population A

* Women without a history of breast cancer and / or ovarian cancer and no family history of breast and / or ovarian cancer among family members on the 1st and 2nd degree before age 50 for breast cancer and before age 60 for ovarian cancer
* Age 18-65 years
* Women targeted for breast reduction surgery
* Agreeing to participate in the study (collection of signed informed consent)

For population B

* Women over the age of 18, with no previous history of breast and / or ovarian cancer and no family history of breast and / or early ovarian cancer in first and second degree relatives, ( diagnosis before age 50 for breast cancer and before age 60 for ovarian cancer).
* Women to be operated on for a hysterectomy with annexectomy or an annexectomy in a benign indication

For population C :

* Women with a history of breast cancer between 50 and 65 years of age but no history of ovarian cancer and no family history of breast and / or ovarian cancer in first- and second-degree relatives before 50 years of age breast cancer and before age 60 for ovarian cancer
* Women who have been treated for breast cancer and undergoing contralateral symmetrization surgery

Exclusion Criteria:

* Men
* Personal history (for population A and B) or family history (populations A, B, C) of breast and / or ovarian cancer (known breast or ovarian cancer in their family of 1st and 2nd degree before age 50 for breast cancer and before age 60 for ovarian cancer)
* Population C: breast cancer under 50 years
* Persons deprived of liberty or guardianship (including curatorship)

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2020-10 (Actual); Study Completion 2020-10 (Actual)

PRIMARY OUTCOMES:
Difference between the average rate of inclusion of exons (exon inclusion mean level) messenger RNA leucocyte of patients and the controls (without matching) | at inclusion

SECONDARY OUTCOMES:
Difference between the average rate of inclusion of exons (exon inclusion mean level) leukocyte messenger RNAs and, the mRNA of breast tissue in healthy women (with pairing). | at inclusion

CONTACTS AND LOCATIONS:
Overall Officials: Sophie KRIEGER, MD, Principal Investigator — Centre François Baclesse
Locations (1):
- Clinique du Parc, Caen, France